CLINICAL TRIAL: NCT07395882
Title: Investigating the Neurophysiology of Itch
Brief Title: A New Model to Induce Itch and Inflammation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N-20250026 Project 1
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Itching
MeSH Terms: conditions — Pruritus | interventions — Histamine; Hot Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active group (Experimental): Heath will be applied prior pruritogens application
  Interventions: Other: Cowhage (Mucuna Pruriens); Other: Histamine; Other: Heat

INTERVENTIONS:
Other: Cowhage (Mucuna Pruriens) — The spicules will be manually inserted. Approximately 30-35 spicules are gently rubbed into a 1 cm diameter skin area on the forearm/face
Other: Histamine — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied
Other: Heat — 45 °C x 5 min

SUMMARY:
This project aims to create a reliable, long-lasting itch model by synergistically combining thermal pre-conditioning with the application of histamine or cowhage.

DETAILED DESCRIPTION:
Two areas (4x4 cm, one on each forearm), will be selected. Initially, superficial blood perfusion will be measured in each area, followed by pruritogens application. During the 10 minutes of the application of the pruritogens, itch will be continuously monitored using a VAS scale. After the pruritogens application, assessment of the superficial blood perfusion (SBP), mechanical sensitivity, and thermal sensitivity will be conducted. The session will be identical to the first session, but pre-heat conditioning will be applied prior to pruritogens application.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g., neuropathy), immunological (e.g., asthma, immune deficiencies, arthritis), musculoskeletal (e.g., muscular pain in the upper extremities), cardiac disorder (e.g., stroke), or psychiatric diagnoses (e.g., depression, bipolar disorders, acute and chronic psychosis) that may affect the results
* Current use of medications that may affect the trial, such as antihistamines, antipsychotics, painkillers, and systemic or topical steroids
* Skin diseases (e.g., atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested (forearm/hand).
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Unable to answer the "Transcranial Magnetic Stimulation Adult Safety Screen" (subprojects 2-4)
* Contraindications to transcranial magnetic stimulation (TMS) application (history of epilepsy, metal implants in head or jaw, etc.) (subprojects 2-4)
* Presence of implanted hearing aids or metal implants on the face, including permanent makeup or tattoos (subprojects 2-4)
* Contraindications to capsaicin, including intolerance to chili or burns or wounds at the application sites (subprojects 2, 3, and 4)
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)
* The subject is assessed as unable to engage in the necessary cooperation required by the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring pain by computerized Visual Analog Scale Scoring | Day 1
  We will ask the subjects to rate the sensation of pain on a 100
Measuring Itch by computerized Visual Analog Scale Scoring | Day 1
  We will ask the subjects to rate the sensation of itch on a 100
Measuring pain by computerized Visual Analog Scale Scoring | Day 2
  We will ask the subjects to rate the sensation of pain on a 100
Measuring Itch by computerized Visual Analog Scale Scoring | Day 2
  We will ask the subjects to rate the sensation of itch on a 100

SECONDARY OUTCOMES:
Superficial blood perfusion | Day 1
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Superficial blood perfusion | Day 2
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Alloknesis | Day 1
  Measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Alloknesis | Day 2
  Measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Mechanically evoked itch (MEI) | Day 1
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanically evoked itch (MEI) | Day 2
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanical Pain Thresholds (MPT) | Day 1
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Thresholds (MPT) | Day 2
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS) | Day 1
  This test is conducted with the same pinprick set used to test the MPT.
Mechanical Pain Sensitivity (MPS) | Day 2
  This test is conducted with the same pinprick set used to test the MPT.
Cold Detection Thresholds (CDT) | Day 1
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Thresholds (CDT) | Day 2
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Day 1
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Day 2
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 1
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 2
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Day 1
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Day 2
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Day 1
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Day 2
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroplasticity and Pain Faculty of Medicine, Aalborg University Selma Lagerløfs Vej 249 9260 Gistrup, Denmark, Aalborg, Aalborg, Denmark